CLINICAL TRIAL: NCT01971255
Title: Evaluation of Anti-Hemagglutinin Antibodies as a Correlate of Protection in an H1N1 Influenza Healthy Human Challenge Model
Brief Title: Evaluation of Anti-Hemagglutinin (Anti-HA) Antibodies as Protection From the Flu in Healthy People
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 130215; 13-I-0215 (Other: United States: The National Institutes of Health)
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Influenza A; HAI; H1N1; Challenge Study; Correlates of Protection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Titer (HAI > or = 1:40) (Experimental): Subjects with prechallenge hemagglutination inhibition (HAI) titers of ≥1:40 were assigned to this group. The human challenge virus, Ca/04/2009/H1N1r Challenge Virus, will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 1 mL of virus will be administered.
  Interventions: Biological: Ca/04/2009/H1N1r Challenge Virus
- Low Titer (HAI < 1:40) (Experimental): Subjects with prechallenge hemagglutination inhibition (HAI) titers of <1:40 were assigned to this group. The human challenge virus, Ca/04/2009/H1N1r Challenge Virus, will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 1 mL of virus will be administered.
  Interventions: Biological: Ca/04/2009/H1N1r Challenge Virus

INTERVENTIONS:
Biological: Ca/04/2009/H1N1r Challenge Virus — The human challenge virus will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 1 mL of virus will be administered.

SUMMARY:
Background:

- Researchers want to know if a certain type of antibody in the blood affects whether people get influenza (the flu). They will study 2 different groups with different levels of anti-HA antibodies and expose them to the flu virus. They will study how the flu develops in a healthy person. This may lead to future studies to develop new vaccines and treatments for the flu.

Objective:

- To study how people can be protected from flu infection.

Eligibility:

- Healthy volunteers 18 to 50 years of age.

Design:

* Participants will be screened through the use of a medical history, physical exam, and laboratory tests.
* Groups of 7 participants will stay in an isolation unit in a hospital for at least 9 days with no visitors.
* Participants will be screened again upon admission. They will also have:
* ECG: soft electrodes will be stuck to the skin. A machine will record the heart s electrical signals.
* Echocardiogram: a small probe will be held to the chest to take pictures of the heart.
* Lung tests: participants will blow into a machine.
* They will also have nasal fluid collected. This will be done either with a swab or with a tube of water washing out the nose. This will be done once every day.
* The flu virus will be sprayed into the participant s nose. This will be done only once.
* Participants will complete a questionnaire on day 1 and twice a day after that for 14 days.
* A medical team will watch participants 24 hours a day. They will go home after 2 days of negative flu tests.
* Participants will have 4 follow-up visits over 8 weeks.

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza, and the threat of new pandemic strains emerging, continues to keep influenza at the forefront of infectious disease and public health research. Mean annual estimates of influenza deaths due to seasonal influenza alone, attributes 36,000 deaths in the US and 250,000 to 500,000 deaths in industrialized countries to influenza. Pandemics can have an even more devastating effect, and we must continue to be prepared by making attempts to reduce the public health impact of this important virus.

Currently, influenza vaccination is the cornerstone of prophylaxis and most effective method available to reduce the impact of influenza on the world s population each year. Data from the 2013 influenza season suggest that current seasonal vaccines held to these standards are greatly underperforming especially in those that really need protection such as the elderly, young, and infirmed.

Multiple factors could play a role in defining the true correlates of protection to influenza infection and disease and many of these factors are yet to be clearly defined. In our own influenza challenge study, protocol 12-I-0077, we have clearly seen evidence that not everyone with a low HAI titer is susceptible to influenza, and that there must be other factors protecting certain individuals. There are many examples like this that demonstrate that there may be much more to immune protection to influenza than just anti-HA antibodies.

Live virus challenge studies have played an important role in defining the correlates of protection of influenza in the past, and we believe they can continue to do so in the future. Since the last time a wild-type influenza challenge has been performed to investigate correlates of protection over 20 years ago, many new scientific tools and a significant increase in knowledge of the immune system have developed. In this study we will enroll participants at different hemagglutinin inhibition titer levels and evaluate this as a correlate of protection to the 2009 H1N1 while exploring the other possible correlates of protection that may be identified. This study represents the first opportunity to examine the correlates of protection of influenza in a fully validated and described wild-type virus challenge model. We believe that studies like this are an ideal use of a wild-type influenza challenge study and can lead to intelligent universal vaccine design as well as a basis to begin evaluating novel vaccine strategies in wild-type challenge studies in the future.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Greater than or equal to 18 and less than or equal to 50 years of age.
2. Agrees to not use tobacco products during participation in this study.
3. Willingness to remain in isolation for the duration of viral shedding (at a minimum 9 days) and to comply with all study requirements.
4. A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

   * Of nonchildbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to and 8 weeks after administration of the influenza challenge virus. Acceptable methods of contraception include 1 or more of the following: 1) male partner who is sterile prior to the female participant s entry into the study and is the sole sexual partner for the female participant; 2) implants of levonorgestrel; 3) injectable progestogen; 4) an intrauterine device with a documented failure rate of < 1%; 5) oral contraceptives; and 6) double barrier methods including diaphragm or condom with a spermicide.
5. Willing to have samples stored for future research.
6. Prechallenge serum hemagglutination inhibition (HAI) titer against the challenge virus of greater than or equal to 1:40 or less than or equal to 1:10 during a screening visit in protocol #11-I-0183
7. HIV uninfected.

EXCLUSION CRITEIRA:

1. Presence of self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Postinfectious or postvaccine neurological sequelae.
2. Have close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons greater than or equal to 65 years of age.
   2. Children less than or equal to 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., asthma).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic metabolic disease (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Individuals who are receiving long-term aspirin therapy.
      * Women who are pregnant or who are trying to become pregnant.
3. Individual with body mass index (BMI) less than or equal to 18.5 and greater than or equal to 40.
4. Smokes more than 4 cigarettes or other tobacco products on weekly basis.
5. Complete blood count (CBC) with differential outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
6. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase, uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
7. Neutropenia below 1,500 cells/mm(3) (Grade 2 or greater)
8. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
9. Clinically significant abnormality on electrocardiogram.
10. Clinically significant abnormality as deemed by the PI on echocardiographic testing.
11. Clinically significant abnormality as deemed by the PI on the Pulmonary Function Test (PFT).
12. Recent acute illness within 1 week of admission to the isolation facility.
13. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
14. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
15. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
16. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
17. Receipt of any non-influenza related unlicensed vaccine within 6 months prior to enrollment.
18. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolites, but not tetrahydrocannabinol (THC) or metabolites).
19. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation
20. Known close contact with anyone known to have influenza in the past 7 days.
21. Any condition or event that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIH data repository BTRIS - Biomedical Translational Research Information System

REFERENCES:
- [Background] Potter CW, Oxford JS. Determinants of immunity to influenza infection in man. Br Med Bull. 1979 Jan;35(1):69-75. doi: 10.1093/oxfordjournals.bmb.a071545. No abstract available. PMID 367490
- [Background] Hobson D, Curry RL, Beare AS, Ward-Gardner A. The role of serum haemagglutination-inhibiting antibody in protection against challenge infection with influenza A2 and B viruses. J Hyg (Lond). 1972 Dec;70(4):767-77. doi: 10.1017/s0022172400022610. PMID 4509641
- [Background] Cox RJ. Correlates of protection to influenza virus, where do we go from here? Hum Vaccin Immunother. 2013 Feb;9(2):405-8. doi: 10.4161/hv.22908. Epub 2013 Jan 4. PMID 23291930
- [Derived] Memoli MJ, Han A, Walters KA, Czajkowski L, Reed S, Athota R, Angela Rosas L, Cervantes-Medina A, Park JK, Morens DM, Kash JC, Taubenberger JK. Influenza A Reinfection in Sequential Human Challenge: Implications for Protective Immunity and "Universal" Vaccine Development. Clin Infect Dis. 2020 Feb 14;70(5):748-753. doi: 10.1093/cid/ciz281. PMID 30953061
- [Derived] Han A, Poon JL, Powers JH 3rd, Leidy NK, Yu R, Memoli MJ. Using the Influenza Patient-reported Outcome (FLU-PRO) diary to evaluate symptoms of influenza viral infection in a healthy human challenge model. BMC Infect Dis. 2018 Jul 28;18(1):353. doi: 10.1186/s12879-018-3220-8. PMID 30055573

RESULTS

PARTICIPANT FLOW:
Groups:
- High Titer (HAI > 1:40): Subjects with prechallenge hemagglutination inhibition (HAI) titers at the time of challenge of =1:40 were assigned to this group.
- Low Titer (HAI < 1:40): Subjects with prechallenge hemagglutination inhibition (HAI) titers at the time of challenge of <1:40 were assigned to this group.
Period: Overall Study
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Started | 32 | 42
Completed | 31 | 40
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- High Titer (HAI > 1:40): Enrolled Subjects with prechallenge hemagglutination inhibition (HAI) titers of =1:40 at the time of planned inoculation were placed in this group.
- Low Titer (HAI < 1:40): Enrolled Subjects with prechallenge hemagglutination inhibition (HAI) titers of <1:40 at the time of planned inoculation and were placed in this group.
- Total: Total of all reporting groups
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40) | Total
Number analyzed (Participants) | 32 | 42 | 74
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 1 | 1
  BTWN | 32 | 41 | 73
  GTE65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 16 | 22 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 4 | 3 | 7
  Not Hispanic or Latino | 27 | 38 | 65
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Hawaiian | 0 | 0 | 0
  Black | 12 | 20 | 32
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Disease Severity Score
Description: This was measured using a validated participant directed questionnaire called FLUPRO. This is then scored daily with a range of score from 0-185. The total score is the sum of all time points the questionnaire is given, which is 16 time points. Therefore the total score range is from 0-2960. 0 would represent no symptoms over the 16 time points while 2960 would represent maximum symptoms and perceived severity at all 16 time points.
Time Frame: Within 28 days after inoculation
Population: The analysis included only those subjects who received the influenza challenge virus and was not found to have a confounding infection (i.e. other respiratory virus infection, urinary tract infection, etc.)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- High Titer (HAI > 1:40): Subjects with prechallenge hemagglutination inhibition (HAI) titers of =1:40 were assigned to this group.
- Low Titer (HAI < 1:40): Subjects with prechallenge hemagglutination inhibition (HAI) titers of <1:40 were assigned to this group.
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
units on a scale | 18 [6 to 34] | 21 [8 to 88]

2. Secondary Outcome: Duration of Shedding (Days)
Description: The number of days total from the time a participant had the first positive test for influenza to their last positive test.
Time Frame: Within 14 days of inoculation
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
Days | 0 [0 to 1] | 2 [1 to 5]

3. Secondary Outcome: Duration of Symptoms (Days)
Description: The number of days a participant experienced any influenza symptoms
Time Frame: within 68 days after inoculation
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
Days | 4 [2 to 5] | 5.5 [3 to 8]

4. Primary Outcome: Number of Patients With Mild to Moderate Influenza Disease (MMID)
Description: This was determined by presence of the combination of symptoms of influenza and presence of a positive clinical test for influenza. If both were present then the participant had positive MMID.
Time Frame: Within 10 days of inoculation
Population: The analysis included only those subjects who received the influenza challenge virus and were not found to have a confounding infection (i.e. other respiratory virus infection, urinary tract infection, etc.) In addition this represents the number of people who were high or low titer at the time of challenge with influenza virus not at screening.
Measure: Number; unit: participants
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
participants | 6 | 29

5. Secondary Outcome: Number of Symptoms
Description: A simple count of the number of unique influenza symptoms the participant experienced.
Time Frame: within 68 days after inoculation
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Number
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
Number | 2 [1 to 4] | 4.5 [2 to 8]

6. Secondary Outcome: Number of Participants With Influenza Symptoms
Description: This was determined by the presence or absence of influenza symptoms.
Time Frame: within 68 days after inoculation
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Number analyzed (Participants) | 25 | 40
participants | 20 | 35

ADVERSE EVENTS:
Arm/Group | High Titer (HAI > 1:40) | Low Titer (HAI < 1:40)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/40
Other Adverse Events (participants affected / at risk) | 10/25 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Titer (HAI > 1:40) (N=25) | Low Titer (HAI < 1:40) (N=40)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Platelet Count Decreased (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase (Investigations) | 2 | 0
Blood sodium increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone abnormal (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No